CLINICAL TRIAL: NCT02951117
Title: A Phase 1b, Open Label, Multicenter, Dose Escalation Study of Venetoclax and ABBV-838 Combination Therapy With Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Venetoclax and ABBV-838 Combination Therapy With Dexamethasone in Participants With Multiple Myeloma Whose Cancer Has Come Back or Had No Response to Recent Cancer Treatment
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-655; 2016-001300-28 (EudraCT Number)
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Multiple Myeloma
Keywords: lymphoid malignancies; Next generation sequencing; Refractory Multiple Myeloma; Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — venetoclax; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A Venetoclax QD + ABBV-838 Q3W + Dexamethasone (Experimental): ABBV-838 administered at cohort-defined doses every 3 weeks (Q3W; starting dose 4.0 mg/kg) in combination with venetoclax (400 mg or 800 mg once daily [QD]) and dexamethasone (40 mg once weekly [Q1W]); once the maximum-tolerated-dose (MTD) and recommended phase two dose (RPTD) are determined, ABBV-838 in combination with venetoclax and dexamethasone at RPTD will be administered in a dose expansion phase of the study.
  Interventions: Drug: Venetoclax; Drug: ABBV-838; Drug: Dexamethasone
- Arm B Venetoclax QD + ABBV-838 Q1W or Q2W + Dexamethasone Q1W (Experimental): Dose escalation portion will investigate either the ABBV-838 weekly (Q1W) or bi-weekly (Q2W) dosing interval in combination with venetoclax (400 or 800 mg QD) and dexamethasone (40 mg Q1W).
  The dose expansion portion will investigate either the ABBV-838 weekly (Q1W) or bi-weekly (Q2W) dosing interval in combination with venetoclax and dexamethasone at the RPTD combination defined from the Dose Escalation portion.
  Interventions: Drug: Venetoclax; Drug: ABBV-838; Drug: Dexamethasone

INTERVENTIONS:
Drug: Venetoclax — Tablet
  Other Names: ABT-199
Drug: ABBV-838 — Intravenous infusion
Drug: Dexamethasone — Tablet or intravenous infusion

SUMMARY:
This is an open-label, multicenter clinical trial designed to evaluate the safety and potential efficacy of venetoclax and ABBV-838 combination therapy with dexamethasone in participants with relapsed or refractory multiple myeloma (MM) who have received 2 or more prior lines of therapy for multiple myeloma (MM). The study will consist of 2 arms: Arm A and Arm B (if applicable). Each arm will have a dose escalation and dose expansion portion.

DETAILED DESCRIPTION:
The study will consist of 2 arms: Arm A and Arm B (if applicable). Arm A dose escalation will investigate up to 3 doses of ABBV-838 at 3-week dosing intervals (Q3W) in combination with venetoclax and dexamethasone. Arm A dose expansion portion will investigate the ABBV-838 Q3W dosing interval with venetoclax and dexamethasone at the recommended phase two dose (RPTD) combination defined from the Dose Escalation portion.

Based on data from the ongoing ABBV-838 monotherapy study (Study M14-467) Arm B dose escalation may be conducted, if deemed necessary. If conducted, Arm B dose excalation will investigate up to 3 doses of ABBV-838 at either weekly (Q1W) or bi-weekly (Q2W) dosing intervals in combination with venetoclax and dexamethasone. Arm B dose expansion portion will investigate either the ABBV-838 Q1W or Q2W dosing interval in combination with venetoclax and dexamethasone at the RPTD combination defined from the Dose Escalation portion.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 for participants in the dose escalation portion of the study and ECOG less than or equal to 2 in the dose expansion portion.
* Received at least 2 prior therapies including an Immunomodulatory Thalidomide Derivative Compounds (IMiD) and a proteasome inhibitor.
* Documented relapsed or progressive multiple myeloma on or after any regimen or is refractory to the most recent line of therapy.
* Received at least 2 prior therapies including an IMiD and a proteasome inhibitor.
* Documented relapsed or progressive multiple myeloma on or after any regimen or is refractory to the most recent line of therapy.
* Eligible for and agree to bone marrow (BM) aspirate prior to treatment start and at designated times per protocol.
* Measurable disease at Screening, defined as at least one of the following M component in serum (greater than or equal to 0.5 g/dL) and/or urine (greater than or equal to 0.2 g excreted in a 24 hour collection sample) or serum free light chain greater than or equal to 100 mg/dL with an abnormal κ/λ ratio of less than 0.26 or greater than 1.65.

Exclusion Criteria:

* Received any anti-myeloma therapy (other than monoclonal antibodies), including chemotherapy, radiotherapy, biological, immunotherapy or an investigational therapy, including targeted small molecule agents within 5 half-lives (or 14 days if half-live unknown) prior to first dose of first dose of venetoclax, ABBV-838, and dexamethasone.
* Received anti-myeloma monoclonal antibodies within 6 weeks prior to first dose of venetoclax, ABBV-838, and dexamethasone.
* Has a significant history of renal, neurologic (peripheral neuropathy), psychiatric, endocrinologic (diabetes mellitus), metabolic, immunologic, cardiovascular, pulmonary or hepatic disease within the last 6 months.
* Received corticosteroid therapy at a dose equivalent to greater than or equal to 4 mg/day of dexamethasone within 3 weeks prior to first dose.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-31 (Estimated); Primary Completion 2020-07-28 (Estimated); Study Completion 2021-04-28 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD), and recommended phase two dose (RPTD) of venetoclax and ABBV-838 combination therapy when administered with dexamethasone | Minimum first cycle of dosing (21 or 28 days, depending on arm)
  The MTD and the RPTD of venetoclax and ABBV-838 combination therapy with dexamethasone will be determined during the dose escalation phase of the study. Once the RPTD combination has been determined, the dose expansion portion will begin.
Number of participants with adverse events | Up to approximately 2 years following the first dose of the last subject enrolled

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of venetoclax | Approximately 43 or 57 days (Treatment Arm A and Treatment Arm B, respectively)
Time to Cmax (Tmax) of venetoclax | Approximately 43 or 57 days (Treatment Arm A and Treatment Arm B, respectively)
Area under the plasma concentration-time curve over the 24-hour dose interval (AUC0-24) of venetoclax | Approximately 43 or 57 days (Treatment Arm A and Treatment Arm B, respectively)
Objective Response Rate (ORR) | Cycle 2 Day 1 and Day 1 of every cycle thereafter for up to 2 years following the first dose of the last subject enrolled
  The Objective Response Rate (ORR) is defined as the proportion of subjects with a response (Stringent Complete Response [sCR], Complete Response [CR], Very Good Partial Response [VGPR] or Partial Response [PR]) based on the International Myeloma Working Group (IMWG) criteria.
Cmax of ABBV-838 | Approximately 43 or 57 days (Treatment Arm A and Treatment Arm B, respectively)
Tmax of ABBV-838 | Approximately 43 or 57 days (Treatment Arm A and Treatment Arm B, respectively)
AUC over the dose interval (AUC0-τ) of ABBV-838 | Approximately 43 or 57 days (Treatment Arm A and Treatment Arm B, respectively)
Total monoclonal anti-CS1 antibody (total mAb) | Approximately 43 or 57 days (Treatment Arm A and Treatment Arm B, respectively)
Monomethyl auristatin E (MMAE) toxin levels | Approximately 43 or 57 days (Treatment Arm A and Treatment Arm B, respectively)
Minimal Residual Disease (MRD) | Cycle 4 Day 1 and treatment completion (up to 2 years following the first dose of the last subject enrolled)
  MRD will be assessed in the bone marrow by next generation sequencing (NGS). MRD negativity in bone marrow aspirates will be defined at 10-5 threshold as assessed by NGS.
Terminal phase elimination rate constant (β) for ABBV-838 | Cycle 1 Day 1
Terminal elimination half-life (t1/2) for ABBV-838 | Cycle 1 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Bueno, MD, Study Director — AbbVie
Locations (3):
- Australia (3):
  - St Vincent´s Hospital /ID# 153022, Darlinghurst
  - St. Vincents Hospital Melbourne /ID# 157925, Fitzroy
  - The Alfred Hospital /ID# 150202, Prahran